CLINICAL TRIAL: NCT00743028
Title: A Single Dose Study Evaluating the Oral Bioavailability and Pharmacokinetics of the Capsule Formulation of ABT-263 in Subjects With Cancer
Brief Title: Assess the Oral Bioavailability of New ABT-263 Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Andrew Krivoshik, MD, PhD, Medical Director, Abbott
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M10-454; NCT00923689 (obsolete NCT alias)
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Lymphocytic Leukemia; Lymphomas; Leukemias
Keywords: Other hematological and non-hematological malignancies
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Leukemia | interventions — navitoclax

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: ABT-263
- 2 (Experimental)
  Interventions: Drug: ABT-263
- 3 (Experimental)
  Interventions: Drug: ABT-263
- 4 (Experimental)
  Interventions: Drug: ABT-263
- 5 (Experimental)
  Interventions: Drug: ABT-263
- 6 (Experimental)
  Interventions: Drug: ABT-263

INTERVENTIONS:
Drug: ABT-263 — Single dose of the current ABT-263 formulation being assessed in ongoing Phase 1/2 studies vs. a single dose of one of the new ABT-263 formulation
  Arms: 1; 2
Drug: ABT-263 — Single dose of the current ABT-263 formulation being assessed in ongoing Phase 1/2a studies vs. a single dose of a new ABT-263 formulation followed by QD dosing with a new ABT-263 formulation for 7 days.
  Arms: 3; 4
Drug: ABT-263 — Single dose of the current ABT-263 formulation being assessed in ongoing Phase 1/2a studies vs. a single dose of a new ABT-263 formulation followed by QD dosing with a new ABT-263 formulation for 7 days.
  Arms: 5; 6

SUMMARY:
This is a randomized, open-label, multicenter crossover study to determine the oral bioavailability of new ABT-263 formulations relative to that of the current ABT-263 formulation being administered in ongoing Phase 1/2a studies. Approximately 36 evaluable subjects with lymphoid malignancies, including chronic lymphocytic leukemia, and solid tumors will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* > or =18 years of age;
* Non-hematologic malignancy or hematologic malignancy that is either relapsed or refractory to standard therapy, or failed up to 5 prior standard therapies or no know effective therapy exists;
* Life expectancy is at least 90 days;
* If clinically indicated, (e.g., subjects over the age of 70) subjects must have documented brain imaging (MRI or CT) negative for subdural or epidural hematoma within 28 days prior to the 1st dose of study drug;
* ECOG performance score of < or = 1;
* Adequate bone marrow, renal and hepatic function per local laboratory reference range as follows:

  * ANC > or = 1,000/µl;
  * Platelets > or = 100,000/mm3;
  * Hemoglobin > or = 9.0 g/dL;
  * serum creatinine < or = 2.0 mg/dL or calculated creatinine clearance > or = 50;
* AST and ALT < or = 3.0 x ULN; Bilirubin < or = 1.5 x ULN. Gilbert's Syndrome may have a Bilirubin > 1.5 x ULN;
* aPTT, PT not to exceed 1.2 x ULN;
* Females must be surgically sterile, postmenopausal, have negative pregnancy test at screening;
* Females not surgically sterile or postmenopausal & non-vasectomized males must practice at least one of the following methods of birth control:

  * Total abstinence from sexual intercourse (minimum one complete menstrual cycle prior to starting study drug);
  * Vasectomized partner;
  * Hormonal contraceptives for at least 3 months prior to study;
  * Double-barrier method (including condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream).

Exclusion Criteria:

* History of/clinically suspicious for cancer-related CNS disease; An allogeneic stem cell transplant.
* Underlying, predisposing condition of bleeding/currently exhibits signs of bleeding.
* History of non-chemotherapy induced thrombocytopenic associated bleeding w/i 1 year prior to the 1st dose.
* Peptic ulcer disease or other hemorrhagic esophagitis/gastritis.
* Active ITP/ history of being refractory to platelet transfusions.
* Significant history of cardiac, renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic/hepatic disease.
* Females pregnant or breast-feeding.
* History of or active medical condition(s) that affects absorption or motility.
* Positive for HIV.
* Other clinically significant uncontrolled condition(s) including, but not limited to: active systemic fungal infection; neutropenic fever w/i 1 wk prior to study drug.
* Steroid therapy w/i 7 days prior to 1st dose for anti-cancer intent.
* Anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal (except hormones for hypothyroidism or ERT)/agonists required to suppress serum testosterone levels [e.g. LHRH, GnRH], any investigational therapy w/i 14 days prior to first dose of study drug.
* Biologic agent w/i 30 days prior to 1st dose.
* Anticoagulation therapy/drugs/herbal supplements affecting platelet function.
* Aspirin w/i 7 days prior to 1st dose.
* Grapefruit/grapefruit products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Assess the oral bioavailability of a new ABT-263 formulation relative to that of the current ABT-263 formulation being assessed in ongoing Phase 1/2a studies. | Two Period crossover design.
Assess the oral bioavailability of a new ABT-263 formulation relative to that of the current ABT-263 formulation being assessed in ongoing Phase 1/2a studies and assess new ABT-263 formulations after once daily dosing (QD) and twice daily dosing (BID). | Three Period crossover design.

SECONDARY OUTCOMES:
Safety measures include number and percentage of subjects having treatment-emergent adverse events tabulated by MedDRA system organ class and preferred term, laboratory test results, lymphocyte enumeration results, vital signs, etc. | Two and three period crossover design

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Site Reference ID/Investigator# 10281, Encinitas, California
  - Site Reference ID/Investigator# 10282, Santa Monica, California
  - Site Reference ID/Investigator# 16341, Bethesda, Maryland
  - Site Reference ID/Investigator# 9441, Lebanon, New Hampshire
  - Site Reference ID/Investigator# 20041, Hackensack, New Jersey